CLINICAL TRIAL: NCT05894330
Title: Perception About Upper Limb Functional Recovery, Barriers & Use of Training Devices Among Stroke Survivors- A Cross-Sectional Survey
Brief Title: Perception About Upper Limb Functional Recovery, Barriers & Use of Training Devices Among Indian Stroke Survivors.
Status: Completed | Type: Observational
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nawaj Pathan, Nawaj Pathan and Sampada Kamlakar, Mahatma Gandhi Mission Institute of Health Sciences
Other Study IDs: MGM-ECRHS/2021/39
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Middle Cerebral Artery With Infarction, Rehabilitation, Upper Limb Recovery, Economic Burdon
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate perceptions regarding affected arm and hand function and their willingness to use devices to enhance upper limb functions among stroke survivors. The main question[s] it aims to answer are:

* what will the stroke survivor's perception of interventions and device development in his/her arm recovery?
* Wheather he is willing to use it for his arm recovery?

DETAILED DESCRIPTION:
Individuals with stroke will be recruited from MGM Hospital and other hospitals from Aurangabad. Participants will be adults (age >30) with stroke and with the capacity to provide written or verbal informed consent, and the ability to communicate verbally/online/phone. Participants will be contacted via phone or email by a member of the research team. If needed personal interviews of the patients will be taken. The research team will consist of the author and one helper Physical Therapy student and the guide. All team members participating in the training will ensure consistency in communications with participants. All the participants will be provided with information about the study objectives and procedures and will be asked if they are willing to participate. If they consent, they will be given one of three options:

1. Complete the survey via phone immediately
2. Complete the survey online. In this case, they will be sent a link to their email to complete an online survey.
3. Complete the survey via personal interview

ELIGIBILITY:
* Inclusion Criteria:
* First-ever stroke
* All stages of stroke
* Onset of a stroke at least 1 year ago
* Age group: 30 to 75
* Both genders included
* Patients diagnosed with MCA (Middle Cerebral Artery) stroke
* Exclusion Criteria:
* Aphasia
* Patients who are unable to follow commands
* Patients with other neurological disorders such as Multiple sclerosis and Parkinson's disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Survivors
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Self Structured Marathi language translated Version Questionnaire | One Month
  It's a 69 item questionnaire to obtain the responses from the stroke survivors about their Upper limb recovery and use of devices for the same. The Obtained responses will be used for the analyze the willingness of stroke clients for use of devices for his/her upper limb arm recovery

CONTACTS AND LOCATIONS:
Locations (1):
- MGM's Institute of Physiotherapy, Aurangabad, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
If requested by genuine researchers or by the university officials through official email communications only.